CLINICAL TRIAL: NCT02359123
Title: Cannabics Capsules as Treatment to Improve Cancer Related Cachexia and Anorexia Syndrome in Advanced Cancer Patients- Pilot Study
Brief Title: Cannabics Capsules as Treatment to Improve Cancer Related CACS in Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cannabics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNBX-001
Record Dates: First submitted 2015-01-26; First posted 2015-02-09 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Cancer Cachexia; Atypical Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cannabics 5mg (Experimental): Patients will be treated initially for 3-4 days with 1x5mg Cannabics capsules per day for gradual adaptation. From the 5th day, patients will be treated 2x5mg capsules per 24 hours for a period of 3 months. However, since some patients may suffer from side effects mainly, dizziness and or anxiety, dosage for these patients will be reduced to 5mg per day.
  Interventions: Other: Cannabics capsules

INTERVENTIONS:
Other: Cannabics capsules — Cannabis extract in an oil formulation
  Other Names: Cannabics SR

SUMMARY:
The main purpose in the treatment of patients with advanced cancer and cancer anorexia cachexia syndrome (CACS) is to prolong life and to improve quality of life (QoL) as far as possible. QoL in patients with CACS is directly related to loss of appetite and loss of weight. Cannabis pills are given in Israel to advanced cancer patients with various symptoms in order to improve their QoL. There is data on safety/toxicity of cannabis, and these pills are given under the regulations of the Israel Ministry of Health.

The purpose of this study is to examine the influence of Cannabics capsules on improving loss of appetite and loss of weight.

DETAILED DESCRIPTION:
Cannabis has long been suggested to stimulate appetite, decrease nausea and vomiting, and improve quality of life in cancer patients. Studies on the efficacy of cannabis for improving CACS and S-NIS have had mixed results. After trials showing improvement in weight gain among AIDS patients, cannabinoids were tested on cancer patients as well. In a controlled, random study comparing dronabinol to a placebo among cancer patients, dronabinol was associated with increased appetite in 38% vs 8% for placebo, and decreased nausea in 20% vs 7%, using acceptable measurement scales. Of the dronabinol patients, 22% gained ≥2 kg, compared with 10.5% of placebo recipients, but this datum did not reach significance, perhaps due to the advanced stage of cancer and the high mortality in both placebo and experimental group (30).

Another randomized study compared dronabinol to megestrol acetate or both treatments together. The research included 469 advanced cancer patients who had been suffering from a substantial appetite loss. A greater percentage of megestrol acetate-treated patients reported appetite improvement compared with dronabinol-treated patients, 75% vs 49% (p=0.0001). Combination treatment resulted in no significant differences compared with megestrol acetate alone. Another study, which included 243 patients, compared the administration of a combination of tetrahydrocannabinol and cannabinol to tetrahydrocannabinol alone, compared to placebo. It should be noted that cannabinoid dosages in the study were low, even in comparison to other studies. No significant differences between the groups were seen regarding improvement in appetite or weight-gain. In these two studies, no substantial side effects of cannabis products were found compared to the other arms. This may be related to the dosages of the drugs given.

A more recent study demonstrated improved chemosensory perception, appetite, sleep, and macronutrient preference in advanced cancer patients. However, the study included less than 50 patients. This research showed improvement in taste and smell perception in patients receiving chemotherapy, as well as appetite and caloric intake in the arm that received dronabinol compared to placebo.

Assessment: Base-line assessment

1. Physician anamnesis and physical examination
2. Complete blood cell count (CBC) and biochemistry test: electrolytes, renal and liver function tests, albumin level, total cholesterol level
3. Blood test for TNF-alpha level
4. Nutrition evaluation, including daily caloric calculation (by using 3 day food diary) and weighting the patient
5. QoL assessment by EORTC C30 and Anorexia/Cachexia Therapy assessment by FAACT questionnaire
6. Evaluation of muscle strength by using hand dynamometer as estimation for muscle mass.

Treatment assessment

1. Physician anamnesis including toxicity assessment according to CTCAE recommendations for acute toxicity, and physical examination including weighing the patient every two weeks in the first month, every month in the coming two months, and every six weeks in the next three months
2. CBC, biochemistry blood test, TNF-alpha level on day 1, and after three months
3. Nutritional intake evaluation on the first week and after three months, based on daily caloric calculation of three day food diary
4. Muscle strength evaluation on day 1 and after three months
5. QOL assessment by EORTC C30 and Anorexia/Cachexia Therapy assessment by FAACT questionnaire on day 1 and after three and six months
6. Safety assessment for early psychiatric side-effects by the Community Assessment of Psychic Experiences (CAPE) questionnaire on day 1 and after 2 weeks and after 3 months.
7. Urine THC- levels one day 1, 2 weeks, 3 months.

Quality-of-Life (QOL) Assessment

QOL will be assessed using the European Organization of Research and Treatment of Cancer core questions on the Quality of Life Questionnaire, version 2 (QLQ-C30) (43) and the Anorexia/Cachexia Therapy (FAACT) questionnaire (44).

Nutrition assessment

1. Daily caloric calculation will be based on the three day food diary. On day 1, the patient will meet the dietitian and receive guidance and instruction of how to complete the diary. The cannabis pills will be given on day 4, after bringing back the three day diary. After three months, the patient will again do a three day food diary and caloric calculation will be made.
2. The caloric calculation will be made with the Ministry of Health Computer software "Zameret".
3. The patient will have telephone support from the dietitian as needed during the days of the diary completion.
4. Cannabics capsules will be given on day 4, after bringing back the three day diary.

Safety assessment:

Community Assessment of Psychic Experiences (CAPE) questionnaire to evaluated possible early psychiatric side-effects will be given in 3 time points, together with measuring the THC level in the urine. Evaluation of other side-effects will be done in every physician visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Histological evidence of an incurable malignancy
3. Estimated life expectancy ≥3 months
4. Performance status ≤2 (ECOG classification)
5. Self-report of weight loss of at least 3kg during the preceding 2 months and/or a dietitian-estimated caloric intake of less than 20 calories/kg of body weight per day
6. Patient believes that loss of appetite or loss of weight is an ongoing problem for him
7. Use of chemotherapy or radiotherapy is permitted
8. Sign of written informed consent

Exclusion Criteria:

1. Ongoing use of tube feedings or parental nutrition
2. Edema or ascites
3. Central nervous system metastases or brain tumors (patients with stable disease in the brain 28 days after treatment can be included in the study)
4. Treatment with adrenal corticosteroids (except for short-term dexamethasone during time of chemotherapy), androgens, progestational agents or other appetite stimulants within the previous two weeks
5. Insulin-requiring diabetes
6. Pregnancy or lactation or unwillingness to use oral contraceptives
7. Other life-threatening medical conditions
8. Anticipated alcohol or barbiturate use during the study period
9. Mechanical obstruction of the alimentary tract, malabsorption, or intractable vomiting
10. Use of cannabis or synthetic cannabinoids in the last four weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
weight gain of ≥10% from baseline weight assessed. | 3 months
  weight gain of ≥10% from baseline weight assessed by weighing the patient every two weeks in the first month, every month in the coming two months, and every six weeks in the next three months

SECONDARY OUTCOMES:
Improvement in appetite | 3 months
  measured by [include analysis, scale, questionnaire, etc.]
Nutritional intake | 3 months
  evaluation on the first week and after three months, based on daily caloric calculation of three day food diary.
Reduction in TNF-alpha | 3 months
  level assessed by CBC, biochemistry blood test, TNF-alpha level on day 1, and after three months
Correlation between THC levels and primary outcome, | 3 months
  assessment by Urine THC- levels one day 1, 2 weeks, 3 months.
QOL will be assessed using the European Organization of Research and Treatment of Cancer core questions on the Quality of Life Questionnaire, version 2 (QLQ-C30) and the Anorexia/Cachexia Therapy (FAACT) questionnaire. | 3 months
  will be assessed using the European Organization of Research and Treatment of Cancer core questions on the Quality of Life Questionnaire, version 2 (QLQ-C30) and the Anorexia/Cachexia Therapy (FAACT) questionnaire.
Safety assessment for early psychiatric side-effects by the Community Assessment of Psychic Experiences | 3 months
  (CAPE) questionnaire on day 1 and after 2 weeks and after 3 months.
Evaluation of muscle strength | 3 months
  using hand dynamometer as estimation for muscle mass on day 1 and after three months.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Bar-Sela, Md, Principal Investigator — Rambam MC
Locations (1):
- Rambam MC, Haifa, Israel

REFERENCES:
- [Derived] Bar-Sela G, Zalman D, Semenysty V, Ballan E. The Effects of Dosage-Controlled Cannabis Capsules on Cancer-Related Cachexia and Anorexia Syndrome in Advanced Cancer Patients: Pilot Study. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419881498. doi: 10.1177/1534735419881498. PMID 31595793